CLINICAL TRIAL: NCT02389764
Title: A Phase II Study of BIBF1120 (Nintedanib) for Patients With Metastatic HER2-Negative Inflammatory Breast Cancer (IBC)
Brief Title: Nintedanib For HER2-Negative Metastatic Inflammatory Breast Cancer (MIBC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0464; NCI-2015-00506 (Other: NCI CTRP)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metastatic inflammatory breast cancer; MIBC; HER2-negative; Breast carcinoma; BIBF 1120; Nintedanib; Phone call
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIBF 1120 (Experimental): Initial dose of BIBF 1120 is 200 mg twice daily orally for a 28 day cycle. Participant called by a member of the study staff every 3 months for up to 1 year after end-of-treatment visit. Participant called by a member of the study staff every 3 months for up to 1 year after end-of-treatment visit.
  Interventions: Drug: BIBF 1120; Behavioral: Phone Call

INTERVENTIONS:
Drug: BIBF 1120 — Initial dose is 200 mg twice daily orally for a 28 day cycle.
  Other Names: Nintedanib
Behavioral: Phone Call — Participant called by a member of the study staff every 3 months for up to 1 year after end-of-treatment visit. These calls should last about 2 minutes.

SUMMARY:
The goal of this clinical research study is to learn if Ofev® (nintedanib, also called BIBF1120) can help to control IBC. The safety of this drug will also be studied.

This is an investigational study. Nintedanib is commercially available and FDA approved for the treatment of certain types of lung disease. Its use in this study is investigational. The study doctor can explain how the study drug is designed to work.

Up to 44 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 4 weeks.

If you are found to be eligible to take part in this study, you will take nintedanib capsules by mouth 2 times each day. Each dose should be about 12 hours apart, at about the same times every day. The capsules should be swallowed whole with about a cup (8 ounces) of water within 30 minutes after eating a meal.

If you forget to take the capsules and it has been more than 2 hours since you were scheduled to take the dose, you should skip that dose and take the next dose as scheduled. Do not double the next dose to "make up" the missed one.

You will be given a study drug diary to write down when you took each dose of study drug. You will need to bring back any empty or partially used bottles of study drug, along with any leftover study drug, with you to the clinic at each cycle.

If you experience side effects, you will be given standard drugs to help decrease the symptoms of the side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

All tests and procedures below will be performed before your dose of study drug.

On Day 1 of every cycle:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.

On Day 1 of Cycles 1-7 and then every odd-numbered cycle after that (Cycles 9,11, 13, and so on), the physical exam and blood draw will be performed at MD Anderson . On Day 1 of Cycles 8 and then every even-numbered cycle after that (Cycles 10, 12, 14, and so on), the physical exam and blood draw may be performed at a local clinic or doctor's office and the results will be sent to the study doctor for review. The study doctor will discuss this option with you.

On Day 1 of Cycle 3, blood (about 2 tablespoons) will also be drawn for biomarker testing.

On Day 1 of Cycles 3, 5, 7, and then every odd numbered cycle after that (Cycles 9, 11, 13, and so on):

* If the doctor thinks it is needed, photographs will be taken of any areas affected by the disease.
* If the doctor thinks it is needed, you will have an x-ray, ultrasound, CT scan, PET/CT scan, and/or a bone scan to check the status of the disease.

At any point that the doctor thinks it is needed, you will have an EKG, ECHO, and/or MUGA scan. You may have any of the above tests/procedures repeated as well, if the doctor thinks it is needed, to check on your health.

Length of Study:

You may continue taking the study drug for up to 2 years. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after you have completed the follow-up period.

End-of-Treatment Visit:

Within 14 days after the last study visit:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, photographs will be taken of your skin and any areas affected by the disease.
* If the doctor thinks it is needed, you will have an x-ray, ultrasound, CT scan, PET/CT scan, and/or a bone scan to check the status of the disease.
* If the doctor thinks it is needed, you will have an EKG and either an ECHO or MUGA scan.

Follow-up Visits:

You will be called by a member of the study staff every 3 months for up to 1 year after your end-of-treatment visit and asked how you are doing. These calls should last about 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are 18 years of age or older
2. Patients are female or male.
3. Have histological confirmation of breast carcinoma with a clinical diagnosis of IBC based on presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast. Pathological evidence of dermal lymphatic invasion should be noted but is not required at diagnosis.
4. Have confirmed distant metastasis with or without local recurrence.
5. Have negative HER2 expression by IHC (defined as 0 or1+), or FISH. If HER2 is 2+, negative HER2 expression must be confirmed by FISH.
6. Patients may undergo an optional biopsy of the metastatic disease at baseline and after 2 cycles of BIBF-1120.
7. Estimated life expectancy of at least 3 months
8. Have ECOG performance status score 0-2
9. Have received at least one any prior treatment for local recurrence or metastatic disease and have relapsed.
10. Signed and dated written informed consent prior to admission to the study
11. If Patients have been treated with anti-VEGF agents, such as Bevacizumab, last dose must be >/= 4 weeks.
12. Have tissues from a biopsy, or have up to 20 unstained slides available from archived metastatic tissue block for biomarker evaluation
13. Patients are able to swallow and retain oral medication

Exclusion Criteria:

1. Patients have an active infection and require IV or oral antibiotics.
2. Patients have impaired cardiac function or clinically significant cardiac diseases, including any of the following: a) History or presence of serious uncontrolled ventricular arrhythmias or presence of atrial fibrillation; b) Clinically significant resting bradycardia (< 50 beats per minute); c) LVEF assessed by 2-D echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) < 45%; d). pericardial effusion
3. Any of the following within 6 months prior to study entry: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF) > NYHA II, Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE),
4. Uncontrolled hypertension defined by an SBP>150 and/or a DBP>100 mm Hg with or without anti-hypertensive medication
5. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug as determined by the investigator.
6. Patients have a concurrent disease or condition that would make them inappropriate for study participation, or any serious medical disorder that would interfere with patients' safety as determined by the investigator.
7. Patients with only locally or regionally confined disease without evidence of metastatic disease
8. Prior treatment with BIBF 1120 or any other VEGFR inhibitor within 4 weeks
9. Known hypersensitivity to the trial drugs , to their excipients or to contrast media
10. Chemotherapy, hormonal therapy, radiotherapy (except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug
11. Persistence of toxicity from previous chemo and/or radiotherapy > grade 2.
12. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomisation).
13. Radiographic evidence of cavitary or necrotic tumors
14. Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
15. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
16. Therapeutic anticoagulation( except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day
17. Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
18. History of clinically significant haemorrhagic or thromboembolic event in the past 6 months
19. Known inherited predisposition to bleeding or thrombosis
20. Proteinuria CTCAE grade 2 or greater
21. Creatinine >/= 1.5 x ULN or GFR < 45 ml/min
22. Hepatic function: total bilirubin outside of normal limits; ALT or AST >1.5 x ULN in pts without liver metastasis. For Pts with liver metastasis: total bilirubin outside of normal limits, ALT or AST >2.5 x ULN
23. Coagulation parameters: International normalised ratio ( INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN
24. Absolute neutrophil count ( ANC) < 1500/ml, platelets < 100000/ml, Haemoglobin < 9.0 g/dl
25. Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix
26. Known history of active or chronic hepatitis C and/or B infection
27. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
28. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females) during the trial and for at least three months after end of active therapy (Contraception in patients with preserved reproductive capacity, patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least two years.)
29. Patients with child bearing potential must have a negative pregnancy test (urine or serum) prior to study treatment
30. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
31. Active alcohol or drug abuse
32. Significant weight loss (> 10% of BW) within past 6 months prior to inclusion into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2019-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was registered twice in error.
Period: Overall Study
Arm/Group | BIBF 1120
Started | 9
Completed | 0
Not Completed | 9
Not completed — Lack of Efficacy | 9

BASELINE CHARACTERISTICS:
Arm/Group | BIBF 1120
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (Complete Response [CR], Partial Response [PR] or Stable Disease [SD] Date) of BIBF 1120 (Nintedanib) in Patients With HER2-negative Metastatic Inflammatory Breast Cancer (IBC).
Description: Clinical benefit defined as participants who achieve CR or PR within 3 months post-treatment, or participants who experience SD for at least three months post-treatment. Clinical benefit rate determined by RECIST 1.1 version." PATHOLOGICAL CR: No evidence of residual invasive tumor, including no residual tumor in the axillary lymph nodes. PR is defined as 30% or greater decrease for a minimum of 4 weeks in the measurable lesion as determined by the product of the perpendicular diameters of the lesion. Every lesion should not regress to qualify as a PR. However, if any lesion progresses or if new lesions appear, the response cannot be classified as a (PR). Minor Response [MR] Decreases in tumor masses insufficient to qualify as a partial remission, i.e. <50%. SD between MR and PD. PD increase in the size by 25% of any measured lesion from baseline. Appearance of new lesions will also constitute increasing disease. Mixed responses will be considered PD.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 9
Participants
  Progressive Disease | 9
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0

2. Secondary Outcome: Safety Measures of BIBF 1120 in Terms of Type, Frequency and Severity of Adverse Event According to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 in Patients With Metastatic IBC.
Description: An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment. All adverse events (grade 3 or higher for hematological toxicity, grade 2 or higher for non-hematological toxicity)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 9
participants
  Grade 3-hematological toxicity | 0
  Grade 4-hematological toxicity | 0
  Grade 2-non-hematological toxicity | 9
  Grade 3-non-hematological toxicity | 4
  Grade 4-non-hematological toxicity | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection was from a complete treatment cycle defined as 28 days or 4 weeks (+/- 2 days) up to 24 months and/or up to 30 days following discontinuation of study drug.
Arm/Group | BIBF 1120
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 (N=9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 (N=9)
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Platelet count decreased (Blood and lymphatic system disorders) | 2
Headache (Nervous system disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Weight loss (Investigations) | 1
Paresthesia (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Shingles (Infections and infestations) | 1
Edema limbs (General disorders) | 1
Hot flashes (Vascular disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT02389764/Prot_SAP_000.pdf